CLINICAL TRIAL: NCT00559663
Title: Flavonoid Effect on Activation and Stimulation of Thrombocytes, hsCRP and Lipid Profile
Acronym: FEAST-CAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LifeBridge Health (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1242; 1242
Record Dates: First submitted 2007-11-15; First posted 2007-11-16 (Estimated); Last update posted 2007-11-20 (Estimated); Status verified 2007-11

CONDITIONS: Healthy
Keywords: Flavonoid; hsCRP; HDL; LDL; platelet reactivity
MeSH Terms: interventions — Tea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GT (Active Comparator): The green tea group is given initially green tea treatment and then after a washout period of four weeks switched to the dark chocolate treatment.
  Interventions: Dietary Supplement: Green tea
- DC (Active Comparator): The dark chocolate group is given initially dark chocolate treatment and then after a washout period of four weeks switched to the green tea treatment.
  Interventions: Dietary Supplement: 70% dark chocolate

INTERVENTIONS:
Dietary Supplement: Green tea — The green tea group consumed first daily one liter of green tea infusate made of 4 bags left in boiling water during 3 minutes.
  After a four week washout-time they were switched over to the dark chocolate treatment, which included consumption of 3.5 ounces 70% dark chocolate.
  Blood was drawn before and after each intervention, to check platelet activity with flow cytometry, HDL, LDL and hsCRP Levels
  Arms: GT
Dietary Supplement: 70% dark chocolate — The dark chocolate group consumed 3.5 ounces 70% dark chocolate per day during a one week period.
  After a four week washout-time they were given the green tea treatment, which included ingestion of one liter green tea infusate (containing 4 green tea bags).
  Blood was drawn before and after each intervention, to check platelet activity with flow cytometry, HDL, LDL and hsCRP Levels.
  Arms: DC

SUMMARY:
The purpose of this study is to compare the effect of dark chocolate with green tea in healthy subjects on clot formation (platelet activity) cholesterol profile and markers of inflammation in two groups.

The first group will be on a regimen of dark chocolate, and the second group will be on a regimen of green tea. Clinical outcomes will be determined after seven days of each treatment and both groups will undergo both treatments subsequently and serve as their own control.

The hypothesis is that both green tea and dark chocolate will reduce platelet activity and reduce LDL, hsCRP and increase HDL.

DETAILED DESCRIPTION:
Flavonoids are polyphenolic compounds ubiquitous in fruits and vegetables. They appear in especially high concentrations in the form of flavanols in green tea as well as in cocoa, and are known to have beneficial antioxidant effects in vitro. Flavonoids have been proposed as a key protective dietary component, reducing the risk of coronary heart disease, including the reduction of elevated blood pressure in persons with hypertension and capable of decreasing LDL.

The aim of this prospective single cross-over study is to assess the effect of green tea and dark chocolate consumption on inhibiting platelet activation, Lipid levels, and hsCRP in healthy volunteers.

This research will be done at Sinai Hospital of Baltimore and will include 35 subjects who will be randomized equally between the two groups.

All blood work will be processed at the Sinai Center for Thrombosis Research. Clinical outcomes will be recorded using a standard case report form.

ELIGIBILITY:
Inclusion Criteria:

* non-smokers between the ages of 18-60
* BMI of 19 to 30

Exclusion Criteria:

* prior usage of Vitamin C > 1000 mg, Vitamin E > 400IU, Beta Carotene > 1000IU, Vitamin A > 5000IU, Selenium > 200mcg, Folic Acid > 1mg, Aspirin or NSAIDs four weeks prior to study initiation
* regular ingestion of Flavonoid rich food (EG green tea, dark chocolate, grapes, red wine and others) prior and during the study except what was provided by the study protocol
* Alcohol or Caffeine consumption 24 prior to blood draws
* Nursing or pregnant women
* blood donation up to eight weeks prior to study initiation
* subjects with coagulation disorders
* known cardiovascular disease (prior myocardial infarction)
* drug abuse
* Diabetes

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2006-09; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
The primary outcome was the absolute change in platelet activity measured by Flow Cytometry, HDL, LDL and hsCRP after dark chocolate, respective green tea treatment. | one week of dark chocolate versus one week of green tea ingestion

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Gurbel, MD, Principal Investigator — Sinai Hospital of Baltimore; Miruais S Hamed, MD, Study Director — Department of Medicine, Sinai Hospital, Baltimore; Kevin Bliden, BS, Study Chair — Sinai Center for Thrombosis Research
Locations (1):
- Center for Thrombosis Research, Sinai Hospital, Baltimore, Maryland, United States